CLINICAL TRIAL: NCT02703727
Title: Durchführung Einer Beobachtungsstudie im Rahmen Einer Masterarbeit Zur Identifikation Von Pharmaceutical Care Issues Bei Patienten, Welche Mit Oralen Antikoagulantien Behandelt Werden
Brief Title: Medication Review Focusing on Anticoagulation Therapy in Swiss Community Pharmacies
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor
Other Study IDs: evalPMC-OAC
Record Dates: First submitted 2016-01-19; First posted 2016-03-09 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Drug Therapy Management
Keywords: polypharmacy; polymedication check; anticoagulation treatment

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OAC: Patients on oral anticoagulation therapy (OAC) will receive a pharmacists led medication review with a focus on anticoagulation therapy (extended polymedication check)
  Interventions: Behavioral: Extended polymedication check

INTERVENTIONS:
Behavioral: Extended polymedication check — Behavioral: Medication review
  Patients on oral anticoagulants and polypharmacy will receive extended polymedication check to identify Pharmaceutical Care Issues, Adherence Issues, Drug related problems and Knowledge Gaps
  The PMC has been implemented in 2010 as a new cognitive service provided by any community pharmacist to patient with polypharmacy (n>3 drugs) on long term conditions (> 3 months) and is reimbursed by swiss health insurance. The semi-structured interview contains questions about knowledge on oral anticoagulation therapy. This extended PMC follows a structured predefined protocol.
  As an outcome, pharmacist may install a compliance support e.g. weekly filled pill organizer.

SUMMARY:
Oral anticoagulation therapy (OAC) entails a high potential for adverse events and strict adherence is needed.Thus, medication review and identification of safety issues and knowledge gaps about OAC is critically important. The polymedication check (PMC) is a reimbursed intermediate medication review focusing on adherence and medication management for Swiss primary care. Investigators aime to assess the impact of the PMC extended with a semi-structured interview focusing on OAC.

ELIGIBILITY:
Inclusion Criteria:

* intake of an oral anticoagulant
* more than 3 drugs over at least 3 months prior to recruitment
* german language (written and spoken)
* medicines use in self management

Exclusion Criteria:

* living in a nursing home
* provision of polymedication check in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with oral anticoagulants (vitamin K antagonists and new oral anticoagulants) on long term polypharmacy ( more than 3 drugs over at least 3 months prior to recruitment) who are able to understand written and oral German language.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of Knowledge gaps about oral anticoagulation therapy | 2 Weeks
  Knowledge about oral anticoagulation therapy will be assessed during the extended Polymedication check which includes 8 specific questions on oral anticoagulation knowledge. After 2 Weeks a follow-up telephone interview will be performed and the same 8 questions will be assessed.

SECONDARY OUTCOMES:
Medication possessio ratio (MPR) | 12 Months
  Medication history from pharmacy software will be used to calculate the MPR of all drugs, retrospectively starting 12 months before the extended PMC takes place.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt E Hersberger, Prof., Principal Investigator — Pharmaceutical Care Research Group
Locations (1):
- Pharmaceutical Care Research Group University of Basel, Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vrijens B, De Geest S, Hughes DA, Przemyslaw K, Demonceau J, Ruppar T, Dobbels F, Fargher E, Morrison V, Lewek P, Matyjaszczyk M, Mshelia C, Clyne W, Aronson JK, Urquhart J; ABC Project Team. A new taxonomy for describing and defining adherence to medications. Br J Clin Pharmacol. 2012 May;73(5):691-705. doi: 10.1111/j.1365-2125.2012.04167.x. PMID 22486599
- [Background] Krska J, Avery AJ; Community Pharmacy Medicines Management Project Evaluation Team. Evaluation of medication reviews conducted by community pharmacists: a quantitative analysis of documented issues and recommendations. Br J Clin Pharmacol. 2008 Mar;65(3):386-96. doi: 10.1111/j.1365-2125.2007.03022.x. Epub 2007 Oct 8. PMID 17922887
- [Background] Clifford S, Barber N, Elliott R, Hartley E, Horne R. Patient-centred advice is effective in improving adherence to medicines. Pharm World Sci. 2006 Jun;28(3):165-70. doi: 10.1007/s11096-006-9026-6. Epub 2006 Sep 27. PMID 17004019
- [Background] Kwint HF, Faber A, Gussekloo J, Bouvy ML. Effects of medication review on drug-related problems in patients using automated drug-dispensing systems: a pragmatic randomized controlled study. Drugs Aging. 2011 Apr 1;28(4):305-14. doi: 10.2165/11586850-000000000-00000. PMID 21428465
- [Background] Bryant LJ, Coster G, Gamble GD, McCormick RN. The General Practitioner-Pharmacist Collaboration (GPPC) study: a randomised controlled trial of clinical medication reviews in community pharmacy. Int J Pharm Pract. 2011 Apr;19(2):94-105. doi: 10.1111/j.2042-7174.2010.00079.x. Epub 2011 Feb 25. PMID 21385240